CLINICAL TRIAL: NCT05078697
Title: Exploratory Study on Gestational Diabetes Mellitus: Multiomics-based Prediction Model
Brief Title: Multiomics-based Prediction Model for GDM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HS-2297
Record Dates: First submitted 2021-09-03; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-05

CONDITIONS: GDM
Keywords: GDM; predictive model; multiotimics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples With DNA — blood, feces, urine, saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- early pregnancy women: According to the 2020 high-risk population score model, participants with high risks for GDM and normal health participants will be enrolled into the study.

SUMMARY:
A prospective cohort study was conducted to :1. explore the relative biomarkers of related with the occurence and development; 2. develop a multiotimics prediction model for GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is one of the most complications during pregnancy and it is associated with many adverse outcomes especially when the pregnant women can't control blood glucose well. With economy develop rapidly, the occurence of GDM is about 15-20%. Recently, the research on GDM has gone into the molecular level, which is beneficial to diagnosis and treatment on GDM. Besides, the cost of hospitalization and treatment for adverse outcomes caused by GDM have caused a certain burden to pregnant women, their families and the whole country. Lifestyle management has the first-line for treatment on GDM, however, the situation of self-management on GDM isn't satisfactory. Therefore, our study aims to explore a model to predict GDM in advance and reduce the adverse outcomes and economy associated with GDM.

The study plan to enroll 60 participants with hisk-risk of GDM and 40 normal participants. They are required sign the inform consent after deciding to participate the research. Furthermore, during early pregnancy (8-13 weeks), middle pregnancy (24-27 3 weeks) and late pregnancy (32-36 weeks), 6-8 weeks after delivery, blood, feces, urine, saliva samples were collected, and continuous blood glucose monitoring system were equipped, human component testing was performed. Follow up was performed to collect the first stool sample of the mother after delivery and faecal samples from the first to the fifth time after birth (the first five times within one week after birth, including hospitalization and discharge) .

ELIGIBILITY:
Inclusion Criteria:

All of following conditions must be met:

* The range of pregnant week is between 8 to 13+6 weeks;
* The range of age is between 20 to 45 years;
* Pregnancy naturally and singleton pregnancy;
* According to the 2020 GDM high-risk population scoring model, those who gets equal to or larger than 80 scores will be assigned to high-risk group and equal to or smaller than 20 scores to low-risk group;

Exclusion Criteria:

Meeting one of the following conditions will be excluded:

* Smoking or drinking alcohols;
* Pregnant women who used antibiotics before 1 month enrollment;
* Combined with Chronic hepatitis, nephritis, chronic gastritis, gastric ulcer, chronic colitis, hyperthyroidism, hypothyroidism (except subclinical hypothyroidism) and blood diseases before pregnancy;
* Pregnant women who has a long-term medication history;
* Those who reject signing the inform consent;
* Those who has participated other clinical trail in the same period

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 60 pregnant women who has high risk for GDM and 40 normal will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
microbiota | At 8 to 13 gestational weeks
  1.The composition of gut and saliva microbiota in women;2. The blood glucose level;3. The body composition value
microbiota | At 24 to 28 gestational weeks
  1.The composition of gut and saliva microbiota in women;2. The blood glucose level;3. The body composition value
microbiota | At 32-36 gestational weeks
  1.The composition of gut and saliva microbiota in women;2. The blood glucose level;3. The body composition value
microbiota | At postpartum 42 days
  1.The composition of gut and saliva microbiota in women;2. The blood glucose level;3. The body composition value; 4. The composition of gut in fetuses

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Chair — Chinese Academic of Medical Science & Peking Union Medical College Hospital
Locations (1):
- Department of ob gyn , Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No